CLINICAL TRIAL: NCT06895382
Title: Comparison of Caudal Epidural Block and Ultrasound-Guided Transversus Abdominis Plane (TAP) Block for Postoperative Analgesia in Pediatric Infraumbilical Surgery: a Randomized Controlled Trial
Brief Title: Caudal Epidural Vs. TAP Block for Postoperative Analgesia in Pediatric Infraumbilical Surgery: a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Onur Baran, Principal Investigator, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TNKU-PED-ANES-2022-001
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain; Pediatric Surgery; Anesthesia, Local; Regional Anesthesia; Abdominal Surgery
Keywords: Caudal Epidural Block; Transversus Abdominis Plane Block; Pediatric Pain Management
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Caudal; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: This study compares two regional anesthesia techniques for postoperative analgesia in pediatric patients undergoing infraumbilical surgery. Participants were randomized into two groups: Group C (Caudal Block) and Group T (TAP Block). Pain scores, analgesic consumption, and adverse effects were compared.
Who Masked: Outcomes Assessor
Masking Description: The study was single-blinded, with postoperative pain assessors blinded to the group allocation. The anesthesiologist administering the block was aware of the group assignment, but postoperative evaluators were not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group C - Caudal Epidural Block (Experimental): Participants in this group received a caudal epidural block after the induction of general anesthesia. A 35-mm 22G or 30-mm 25G block needle was inserted through the sacrococcygeal ligament into the epidural space under aseptic conditions. After confirming negative aspiration for cerebrospinal fluid or blood, 1 mL/kg of 0.25% bupivacaine was administered.
  Interventions: Procedure: Caudal Epidural Block; Drug: Bupivacaine 0.25%
- Group T - Transversus Abdominis Plane (TAP) Block (Experimental): Participants in this group received an ultrasound-guided transversus abdominis plane (TAP) block after the induction of general anesthesia. A 22G, 50-mm insulated block needle was inserted using an in-plane technique under ultrasound guidance with a linear probe. The needle was advanced into the fascial plane between the internal oblique and transversus abdominis muscles. After confirming placement with a 0.5-1 mL test dose of 0.9% NaCl and negative aspiration for blood, 0.3 mL/kg of 0.25% bupivacaine was administered.
  Interventions: Procedure: Transversus Abdominis Plane (TAP) Block; Drug: Bupivacaine 0.25%

INTERVENTIONS:
Procedure: Caudal Epidural Block — A caudal epidural block was performed after the induction of general anesthesia. Using a 35-mm 22G or 30-mm 25G block needle, the sacral hiatus was identified, and the needle was inserted through the sacrococcygeal ligament into the epidural space under aseptic conditions. After confirming negative aspiration for cerebrospinal fluid or blood, 1 mL/kg of 0.25% bupivacaine was administered.
  Other Names: Caudal Block; Caudal Anesthesia
  Arms: Group C - Caudal Epidural Block
Procedure: Transversus Abdominis Plane (TAP) Block — A transversus abdominis plane (TAP) block was performed after the induction of general anesthesia. Using a 22G, 50-mm insulated block needle, the injection was administered under ultrasound guidance using a linear probe and in-plane technique. The needle was advanced into the fascial plane between the internal oblique and transversus abdominis muscles. After confirming placement with a 0.5-1 mL test dose of 0.9% NaCl and negative aspiration for blood, 0.3 mL/kg of 0.25% bupivacaine was administered.
  Other Names: TAP Block; Ultrasound-Guided TAP Block
  Arms: Group T - Transversus Abdominis Plane (TAP) Block
Drug: Bupivacaine 0.25% — 0.25% bupivacaine was administered in both intervention arms as part of the regional anesthesia procedure In the Caudal Block group, 1 mL/kg of 0.25% bupivacaine was administered into the caudal epidural space.
  In the TAP Block group, 0.3 mL/kg of 0.25% bupivacaine was administered into the transversus abdominis plane under ultrasound guidance

SUMMARY:
This randomized controlled trial investigates the postoperative analgesic efficacy of caudal epidural block versus ultrasound-guided transversus abdominis plane (TAP) block in pediatric patients undergoing infraumbilical surgery.

A total of 60 pediatric patients (aged 1 to 7 years, ASA I-II) were randomly assigned to one of two groups:

* Group C (Caudal Block): Received 1 mL/kg of 0.25% bupivacaine in the caudal epidural space.
* Group T (TAP Block): Received 0.3 mL/kg of 0.25% bupivacaine injected into the transversus abdominis plane under ultrasound guidance.

Primary Outcome:

* Postoperative FLACC pain scores at 2, 6, 12, and 24 hours.

Secondary Outcomes:

* Total analgesic consumption (including rescue analgesia).
* Intraoperative hemodynamic parameters (heart rate, blood pressure, SpO₂).
* Incidence of nausea and vomiting (PONV).
* Parental satisfaction scores.

The study aims to determine which regional anesthesia technique provides superior pain relief and reduces systemic analgesic requirements in pediatric patients.

DETAILED DESCRIPTION:
Postoperative pain management in pediatric patients is a challenge due to difficulties in pain assessment and concerns about opioid-related adverse effects. While caudal epidural block has traditionally been the standard of care for infraumbilical pediatric surgeries, ultrasound-guided transversus abdominis plane (TAP) block has emerged as a promising alternative with the potential for longer-lasting analgesia and fewer motor block complications.

This randomized controlled trial was conducted at Tekirdağ Namık Kemal University Hospital between December 2022 and December 2023. A total of 60 pediatric patients (aged 1-7 years, ASA I-II) undergoing infraumbilical surgery were enrolled and randomly assigned to receive either:

* Caudal epidural block (1 mL/kg of 0.25% bupivacaine via the sacral hiatus).
* TAP block (0.3 mL/kg of 0.25% bupivacaine in the fascial plane between the internal oblique and transversus abdominis muscles under ultrasound guidance).

General anesthesia was induced using sevoflurane inhalation, followed by propofol (2-3 mg/kg) and fentanyl (1 µg/kg) for IV induction. A laryngeal mask airway (LMA) was used, and anesthesia was maintained with sevoflurane at a MAC of 1.0%.

Outcome Measures:

* Primary Outcome:

  * FLACC pain scores at 2, 6, 12, and 24 hours postoperatively.
* Secondary Outcomes:

  * Total postoperative analgesic consumption (including rescue analgesia).
  * Hemodynamic parameters (HR, SBP, DBP, SpO₂) recorded at predefined intraoperative time points.
  * Incidence of postoperative nausea and vomiting (PONV).
  * Parental satisfaction scores collected post-discharge.

Statistical Analysis:

Data were analyzed using SPSS 25.0. Sample size was determined using G*Power 3.1.9.2, with an effect size (d) of 0.75, power of 0.80, and Type I error of 0.05. The study followed randomized allocation with blinding of pain assessors.

This study aims to determine whether TAP block provides equivalent or superior analgesia compared to caudal epidural block in pediatric patients undergoing infraumbilical surgeries. Findings will help guide future pediatric regional anesthesia protocols.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 1 to 7 years.
* ASA Physical Status I-II.
* Undergoing infraumbilical abdominal surgery (e.g., hernia repair, orchiopexy, circumcision).
* Parental written informed consent obtained.

Exclusion Criteria:

* Contraindications to regional anesthesia, such as:
* Coagulopathy or bleeding disorders.
* Local infection at the injection site.
* Known allergy to local anesthetics.
* Neurological conditions (e.g., degenerative neuropathy, brain tumors, increased intracranial pressure).
* Intellectual disabilities affecting pain assessment.
* Chronic pain conditions or opioid use before surgery.
* Parental refusal to participate in the study.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Postoperative FLACC Pain Scores | FLACC pain scores were recorded at 2, 6, 12, and 24 hours postoperatively
  Postoperative pain intensity was measured using the Face, Legs, Activity, Cry, Consolability (FLACC) scale at predefined time points after surgery. The FLACC scale is a validated tool for assessing postoperative pain in pediatric patients based on behavioral observations.

SECONDARY OUTCOMES:
Total Postoperative Analgesic Consumption | 0-24 hours postoperatively
  The total amount of rescue analgesia (paracetamol, NSAIDs, opioids) administered in the first 24 hours postoperatively was recorded. This includes any additional medication given based on the patient's pain score.
Intraoperative Hemodynamic Stability | Baseline, after induction, after surgical incision, and at 15, 30, 45, and 60 minutes intraoperatively.
  Heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), and arterial oxygen saturation (SpO₂) were recorded at predefined intraoperative time points to assess the hemodynamic effects of the regional anesthesia techniques.
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-24 hours postoperatively
  The number of patients experiencing postoperative nausea and vomiting (PONV) within the first 24 hours was recorded.
Parental Satisfaction Scores | Recorded at 24 hours postoperatively and at a follow-up phone call after discharge.
  Parental satisfaction with their child's postoperative pain management was assessed using a 5-point Likert scale, ranging from 1 (very dissatisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Onur Baran, Study Chair — Namik Kemal University
Locations (1):
- Tekirdag Namik Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No